CLINICAL TRIAL: NCT04953676
Title: A Randomized, Controlled, Multi-center Clinical Trial of the Round-tunnel and Flat-tunnel Technique of Anterior Cruciate Ligament (ACL) Reconstruction
Brief Title: A Clinical Trial of the Round-tunnel and Flat-tunnel Technique of ACL Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Zhengzhou Orthopaedic Hospital (Unknown); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M2020149
Record Dates: First submitted 2021-06-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): round tunnel
  Interventions: Procedure: round tunnel technique
- Experimental group (Experimental): flat tunnel
  Interventions: Procedure: flat tunnel technique

INTERVENTIONS:
Procedure: round tunnel technique — Both the femoral tunnel and tibial tunnel were drilled by 8-mm cannulated drill
  Arms: Control Group
Procedure: flat tunnel technique — Both the femoral tunnel and tibial tunnel were dimension of 5×11-mm rounded-rectangular, which was created by initially drilling a round tunnel with a 5-mm cannulated drill and reshaped by use of a bone rasp and custom-made dilator.
  Arms: Experimental group

SUMMARY:
This study intends to perform round-tunnel and flat-tunnel ACL reconstruction technique in 144 patients, and compare the clinical outcomes of the two surgical procedures through follow-up.

DETAILED DESCRIPTION:
This is a prospective randomized, controlled, multi-center clinical trial study on ACL reconstruction surgery technique. It is jointly undertaken by the Peking University Third Hospital, Nanjing Drum Tower Hospital, Zhengzhou Orthopaedic Hospital, and Shenzhen Second People's Hospital. Peking University Third Hospital is the team leader unit. In this study, 144 patients with ACL rupture were recruited according to the enrollment criteria. Among them, 54 patients with ACL rupture were recruited and carried out by the Peking University Third Hospital. The recruited patients were randomly divided into groups. The ratio of the control group is 1:1. Each of the other three hospitals recruited 30 patients and randomly grouped them according to the same enrollment criteria. The ratio of the experimental group to the control group was also 1:1. In this study, 72 patients with ACL rupture in the experimental group will be treated with flat-tunnel reconstruction technique, and 72 patients with ACL rupture in the control group will be treated with round-tunnel technique. All operations will be performed with autologous hamstring tendons. After reconstruction, all subjects will participate in the collection of clinical function scores including Tegner score, Lysholm score, IKDC score, and clinical evaluation including physical examination, joint laxity, CT and MRI imaging analysis to verify ACL Advantages of flat-tunnel technique.

ELIGIBILITY:
Inclusion Criteria:

* For the first time, the knee joint simply ruptures the anterior cruciate ligament (ACL) and requires surgical reconstruction; it can be combined with meniscus injury, and the Outerbridge injury score is ≤ Grade II; There is no history of trauma or fracture of the ipsilateral knee joint; Posterior Cruciate Ligament (PCL) has no damage; Medial Collateral Ligament (MCL) or Lateral collateral ligaments (LCL) has no damage or only slight damage (no more than I degree).

Exclusion Criteria:

* BMI is less than 18.5 or greater than 35 kg/m2; Patients with moderate or severe knee degeneration; Those with limited flexion angle (<120 degrees); The cartilage defect area is greater than 2 cm2 or the Outerbridge damage score is> Grade II.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
KT-2000 | 6 months, 12 months, 24 months
  side-to-side difference

SECONDARY OUTCOMES:
Tegner Score | 6 months, 12 months, 24 months
  functional scores
Lysholm Score | 6 months, 12 months, 24 months
  functional scores
IKDC Score | 6 months, 12 months, 24 months
  functional scores
Lachman test | 6 months, 12 months, 24 months
  physical examination
Pivot-shift test | 6 months, 12 months, 24 months
  physical examination

IPD SHARING:
Plan to Share IPD: Undecided